CLINICAL TRIAL: NCT02449980
Title: Primary Versus Delayed Surgical Therapy for Pediatric Spontaneous Pneumothorax: A Randomized Controlled Trial
Brief Title: Primary Versus Delayed Surgical Therapy for Pediatric Spontaneous Pneumothorax
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB recommended termination on the basis of poor accrual rate. We will transition to a prospective observational (non-randomized) study design.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Monica Esperanza Lopez, Associate Professor of Surgery and Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-32402
Record Dates: First submitted 2015-05-12; First posted 2015-05-21 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Pneumothorax
Keywords: Spontaneous Pneumothorax; Video Assisted Thoracoscopic Surgery; Tube Thoracostomy; Pediatric Surgery
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Surgery Group (Active Comparator): Patients randomized to the primary surgical intervention group will undergo VATS (video-assisted thoracoscopic surgery), apical blebectomy and mechanical pleurodesis during the initial hospital admission by the admitting staff surgeon. The general principles of the surgical technique consist of a 3-port thoracoscopic approach, stapled blebectomy, apical mechanical pleurodesis, and placement of chest tube . Variations of this technique will be at the discretion of the surgeon.
  Interventions: Procedure: Primary Surgery Group
- Initial Non-operative management (Active Comparator): Those randomized to the control group will be admitted and their chest tube or percutaneous drainage catheter managed according to standard protocol. This consists of a minimum of 48 hours of Pleur-Evac suction and daily chest radiographs. The drainage tube is then placed to water seal when resolution of the pneumothorax is documented by x-ray, as well as absence of an air leak. If there are no clinical or radiographic changes after a water seal period, the chest tube is then removed. A post-removal chest radiograph is obtained and the patient is discharged if clinical and radiographic criteria are met.
  Interventions: Procedure: Initial Non-operative management

INTERVENTIONS:
Procedure: Primary Surgery Group — Patients will receive surgical intervention during the initial hospital admission, as previously described, for the spontaneous pneumothorax. Patients will then be admitted postoperatively and monitored until discharge criteria are met
  Arms: Primary Surgery Group
Procedure: Initial Non-operative management — Patients will receive percutaneous drainage or chest tube placement as initial management for spontaneous pneumothorax. This will be followed by an observation period until discharge criteria are met.
  Arms: Initial Non-operative management

SUMMARY:
The purpose of this study is to compare the effectiveness of two treatment strategies--delayed versus immediate surgery-- for children with primary spontaneous pneumothorax (collapse of the lung). Currently, both treatment modalities are used and there is no clear evidence that either option is superior. The investigators hypothesize that immediate surgery will have better outcomes with lower recurrence rates than delayed surgery.

DETAILED DESCRIPTION:
1. All children presenting to Texas Children's Hospital with a primary spontaneous pneumothorax will be potentially eligible for the study.
2. After the diagnosis has been made and initial medical therapy has been initiated, the patients will be identified and parents or legal guardian approached by the staff surgeon for consent to participate in the study. The attending pediatric surgeon or surgical fellow will discuss the trial with all eligible patients and their families.
3. Written, informed consent will be obtained by the research nurse coordinator, a pediatric surgical fellow, or an attending pediatric surgeon.
4. Once enrolled, the patients will be randomized to primary surgery: Video-Assisted Thoracoscopic Surgery (VATS), blebectomy and mechanical pleurodesis, versus initial nonoperative treatment.
5. Prior to initiating the study, the randomization sequence will be computer-generated by an independent statistician using a permuted block random allocation scheme with a block size of 4,6. The randomization sequence will be maintained securely within the randomization module in REDCap (Research electronic data capture), and it will be accessed only after enrollment has occurred and inclusion criteria are verified by the admitting staff surgeon. The participants and the surgeons will not be blinded to group assignment.
6. Primary Surgery Group. Patients randomized to the primary surgical intervention group will undergo VATS, apical blebectomy and mechanical pleurodesis during the initial hospital admission by the admitting staff surgeon. The general principles of the surgical technique consist of a 3-port thoracoscopic approach, stapled blebectomy, apical mechanical pleurodesis, and placement of chest tube . Variations of this technique will be at the discretion of the surgeon.
7. Initial non-operative management group. Those randomized to the control group will be admitted and their chest tube or percutaneous drainage catheter managed according to standard protocol. This consists of a minimum of 48 hours of Pleur-Evac suction and daily chest radiographs. The drainage tube is then placed to water seal when resolution of the pneumothorax is documented by x-ray, as well as absence of an air leak. If there are no clinical or radiographic changes after a water seal period, the chest tube is then removed. A post-removal chest radiograph is obtained and the patient is discharged if clinical and radiographic criteria are met. "Rescue" VATS/ blebectomy/pleurodesis will be performed in those managed initially nonoperatively who meet criteria for surgery thereafter (i.e. develop a persistent air leak after drainage tube placement). A persistent air leak will be defined as bubbling of air in the Pleur-Evac water chamber upon eliciting positive pressure lasting >4 days, noted and documented in progress note by attending physician. If recurrence is identified in the control group, it will be managed operatively, as per current clinical practice, with VATS/ blebectomy/pleurodesis.
8. Discharge Criteria. Discharge criteria include being afebrile for 24 hours, normal oxygen saturation with no oxygen requirement, benign physical exam, unchanged or improved post-removal chest radiograph, ability to tolerate regular diet and ambulate, and pain well controlled on oral pain medication.
9. Discharge Instructions. A discussion will take place between the surgical team and the family prior to discharge in order to review standardized discharge instructions. These will address an understanding by the patient and family of the signs and symptoms of recurrent pneumothorax as well as specific follow up appointments and the scheduled phone follow-up thereafter. For patients who have had primary surgery, specific postoperative instructions will be given according to current clinical practice.
10. Follow-up. Follow-up will be the same for both groups and will take place at 2-3 weeks after hospital discharge (per standard of care), with subsequent telephone interviews at 3 months, 6 months and 12 months.
11. The primary outcome regarding effectiveness of primary VATS will be the overall recurrence rate at 12 months. Secondary outcomes include surgical complication rate, cumulative hospital length of stay (total number of hospital days during study period), time to resumption of usual activities, and direct variable hospital costs. The recurrence rate is defined as the proportion of patients with recurrent ipsilateral pneumothorax during the follow-up period. Complications to be assessed include surgical site infection, persistent air leak (> 4 days), and prolonged need for chest tube (as quantified by number of chest tube days). Standard National Surgical Quality Improvement Program (NSQIP) definitions of these outcomes will be utilized. The time to resumption of usual activities will be adjudicated at the time of the post-op follow up visit or by means of a phone interview at 2-3 weeks postoperatively. The longest time period to resumption all usual activities will be ascertained from patient questionnaires addressing return to school date, level of pre- and post-illness activity, and daily activity log kept by the patient or their parent. Post-operative quality of life will be assessed at 3 months, 6 months, and 12 months by telephone administration of The PedsQL Measurement Model for the Pediatric Quality of Life Inventory, a widely-used and validated tool.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 5 to 18 with clinical diagnosis of primary spontaneous pneumothorax (symptoms of chest pain and/or shortness of breath and pneumothorax demonstrated on chest radiograph) and no prior history of pneumothorax

Exclusion Criteria:

* Blunt or penetrating trauma
* Cystic fibrosis
* Pneumonia
* Uncontrolled asthma with hospitalization for exacerbation within previous 30 days
* Congenital cystic adenomatoid malformation or congenital lobar emphysema
* History of previous cardiac or pulmonary surgery

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | 1 month
  The recurrence rate is defined as the proportion of patients with recurrent ipsilateral pneumothorax during the follow-up period.
Recurrence rate | 3 months
  The recurrence rate is defined as the proportion of patients with recurrent ipsilateral pneumothorax during the follow-up period.
Recurrence rate | 6 months
  The recurrence rate is defined as the proportion of patients with recurrent ipsilateral pneumothorax during the follow-up period.
Recurrence rate | 12 months

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Surgical site infection (NSQIP definition), persistent air leak (> 4 days), and prolonged need for chest tube (as quantified by number of chest tube days)
Hospital Length of stay | 1 month
Time to return to normal activities | 1 month, 3 months, 6 months, 12 months
Hospital Direct Variable Costs (in US dollars, from hospital cost-accounting department) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Monica E Lopez, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Sahn SA, Heffner JE. Spontaneous pneumothorax. N Engl J Med. 2000 Mar 23;342(12):868-74. doi: 10.1056/NEJM200003233421207. No abstract available. PMID 10727592
- [Background] Dotson K, Timm N, Gittelman M. Is spontaneous pneumothorax really a pediatric problem? A national perspective. Pediatr Emerg Care. 2012 Apr;28(4):340-4. doi: 10.1097/PEC.0b013e31824d9a65. PMID 22453728
- [Background] Robinson PD, Cooper P, Ranganathan SC. Evidence-based management of paediatric primary spontaneous pneumothorax. Paediatr Respir Rev. 2009 Sep;10(3):110-7; quiz 117. doi: 10.1016/j.prrv.2008.12.003. Epub 2009 May 21. PMID 19651381
- [Background] O'Lone E, Elphick HE, Robinson PJ. Spontaneous pneumothorax in children: when is invasive treatment indicated? Pediatr Pulmonol. 2008 Jan;43(1):41-6. doi: 10.1002/ppul.20734. PMID 18041754
- [Background] Waller DA, Forty J, Morritt GN. Video-assisted thoracoscopic surgery versus thoracotomy for spontaneous pneumothorax. Ann Thorac Surg. 1994 Aug;58(2):372-6; discussion 376-7. doi: 10.1016/0003-4975(94)92210-1. PMID 8067834
- [Background] Kim J, Kim K, Shim YM, Chang WI, Park KH, Jun TG, Park PW, Chae H, Lee KS. Video-assisted thoracic surgery as a primary therapy for primary spontaneous pneumothorax. Decision making by the guideline of high-resolution computed tomography. Surg Endosc. 1998 Nov;12(11):1290-3. doi: 10.1007/s004649900842. PMID 9788848
- [Background] Donahue DM, Wright CD, Viale G, Mathisen DJ. Resection of pulmonary blebs and pleurodesis for spontaneous pneumothorax. Chest. 1993 Dec;104(6):1767-9. doi: 10.1378/chest.104.6.1767. PMID 8252960
- [Background] Cook CH, Melvin WS, Groner JI, Allen E, King DR. A cost-effective thoracoscopic treatment strategy for pediatric spontaneous pneumothorax. Surg Endosc. 1999 Dec;13(12):1208-10. doi: 10.1007/pl00009622. PMID 10594267
- [Background] Poenaru D, Yazbeck S, Murphy S. Primary spontaneous pneumothorax in children. J Pediatr Surg. 1994 Sep;29(9):1183-5. doi: 10.1016/0022-3468(94)90795-1. PMID 7807340
- [Background] Butterworth SA, Blair GK, LeBlanc JG, Skarsgard ED. An open and shut case for early VATS treatment of primary spontaneous pneumothorax in children. Can J Surg. 2007 Jun;50(3):171-4. PMID 17568487
- [Background] Seguier-Lipszyc E, Elizur A, Klin B, Vaiman M, Lotan G. Management of primary spontaneous pneumothorax in children. Clin Pediatr (Phila). 2011 Sep;50(9):797-802. doi: 10.1177/0009922811404699. Epub 2011 Apr 11. PMID 21482575
- [Background] Qureshi FG, Sandulache VC, Richardson W, Ergun O, Ford HR, Hackam DJ. Primary vs delayed surgery for spontaneous pneumothorax in children: which is better? J Pediatr Surg. 2005 Jan;40(1):166-9. doi: 10.1016/j.jpedsurg.2004.09.042. PMID 15868579
- [Background] Baumann MH, Strange C, Heffner JE, Light R, Kirby TJ, Klein J, Luketich JD, Panacek EA, Sahn SA; AACP Pneumothorax Consensus Group. Management of spontaneous pneumothorax: an American College of Chest Physicians Delphi consensus statement. Chest. 2001 Feb;119(2):590-602. doi: 10.1378/chest.119.2.590. PMID 11171742
- [Background] MacDuff A, Arnold A, Harvey J; BTS Pleural Disease Guideline Group. Management of spontaneous pneumothorax: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii18-31. doi: 10.1136/thx.2010.136986. No abstract available. PMID 20696690
- [Background] Ozcan C, McGahren ED, Rodgers BM. Thoracoscopic treatment of spontaneous pneumothorax in children. J Pediatr Surg. 2003 Oct;38(10):1459-64. doi: 10.1016/s0022-3468(03)00496-2. PMID 14577068
- [Background] Cardillo G, Facciolo F, Giunti R, Gasparri R, Lopergolo M, Orsetti R, Martelli M. Videothoracoscopic treatment of primary spontaneous pneumothorax: a 6-year experience. Ann Thorac Surg. 2000 Feb;69(2):357-61; discussion 361-2. doi: 10.1016/s0003-4975(99)01299-0. PMID 10735663
- [Background] Tunis SR, Stryer DB, Clancy CM. Practical clinical trials: increasing the value of clinical research for decision making in clinical and health policy. JAMA. 2003 Sep 24;290(12):1624-32. doi: 10.1001/jama.290.12.1624. PMID 14506122